CLINICAL TRIAL: NCT05102188
Title: Addressing Health Disparities in African Americans - Exploring Sleep and Developing Interventions -2
Brief Title: Addressing Health Disparities in African Americans - Exploring Sleep and Developing Interventions - 2
Acronym: HD-SLEEP2
Status: Completed | Type: Observational
Sponsor: Pennington Biomedical Research Center (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Principal Investigator, Prachi Singh, Associate Professor, Sleep and Cardiometabolic Health, Pennington Biomedical Research Center
Other Study IDs: PBRC 2020-020-2; U54GM104940 (NIH)
Record Dates: First submitted 2021-10-20; First posted 2021-11-01 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Sleep
Keywords: African American; Sleep

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- African American adults with poor sleep: Individuals with self-identified poor sleep quality and/or quantity
  Interventions: Combination Product: Assessment of sleep and related factors

INTERVENTIONS:
Combination Product: Assessment of sleep and related factors — Eligible participants will be invited to fill out several forms and wear a watch-like device on their wrist (an accelerometer) for 7 days to assess their sleep habits. They will also be asked to sleep at home with a watch-like device attached to a sleeve which covers their index finger (an oximeter) for one night to assess whether they may have a sleep problem like sleep apnea.

SUMMARY:
The purpose of the HD-SLEEP2 study is to help researchers understand sleep in African Americans. The investigators also want to know what factors may affect sleep.

DETAILED DESCRIPTION:
African Americans who self-report poor sleep (n=80) will be invited to complete questionnaire based self-assessment of known factors and comorbidities contributing to alterations in sleep such as demographic characteristics, anthropometrics, depression, insomnia, and food habits in conjunction with objective and subjective measures of sleep via 7-day accelerometry (sleep duration), overnight oximetry (sleep apnea), and sleep questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Self-identified African American
* Age range: >18 years (inclusive)
* Sex: Both males and females will be allowed to participate in the study
* Self-perceived poor sleep

Exclusion Criteria:

* Unable to provide written informed consent
* Unable to understand English

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: African Americans residing in Greater Baton Rouge area will be invited to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2022-03-11 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Habitual sleep duration | 7 days
  Average hours of sleep/24h period
Oxygen desaturation index | 1 day
  Number of oxygen desaturation events per hour of sleep
Sleep Quality | 1 day
  Sleep quality as determined by Pittsburgh Sleep Quality Index. The minimum score is 0 and maximum score is 21. Higher scores indicate poor sleep quality.
Daytime Sleepiness | 1 day
  Severity of daytime sleepiness as determined by Epworth Sleepiness scale. The minimum score is 0 and maximum score is 24. Higher scores suggest daytime sleepiness.
Sleep behaviors | 1 day
  Sleep hygiene behaviors as determined by sleep hygiene index. The minimum score is 13 and maximum score is 65. Higher scores indicate poor sleep hygiene status.

CONTACTS AND LOCATIONS:
Overall Officials: Prachi Singh, PhD, Principal Investigator — Pennington Biomedical Research Center
Locations (1):
- Recruiting core Pennington, Baton Rouge, Louisiana, United States

IPD SHARING:
Plan to Share IPD: Undecided